CLINICAL TRIAL: NCT00184418
Title: The Immune System and Psychiatric Disorders
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 94463
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Stress Disorders, Traumatic; Depressive Disorder; Bipolar Disorder; Personality Disorders; Schizophrenia; Psychotic Disorders
Keywords: Immunity; Immune System; Cytokines; Psychophysiology; Psychoneuroimmunology
MeSH Terms: conditions — Stress Disorders, Traumatic; Depressive Disorder; Bipolar Disorder; Personality Disorders; Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, frozen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients admitted to a psychiatric acute ward

SUMMARY:
The study is based on a hypothesis that there is interaction between the activity in the immune system and in the mind. To study this, the investigators register different measures for activity in the immune system on patients unselectedly admitted to an acute psychiatric ward. The psychiatric statuses and diagnoses of these patients are carefully defined as well.

DETAILED DESCRIPTION:
Our hypotheses are first that activity in the immune system influences the psychiatric status in general, second that changes in activity in psychiatric status affect activity in the immune system and third that there are connections between certain psychiatric conditions/disorders and certain features of the immune system.

All patients admitted to a psychiatric acute ward covering an area with a population of 130.000 and with around 1000 admittances to an acute psychiatric ward a year (some readmittances) are asked to participate in the study. Patients fill in a question form regarding psychiatric as well as somatic health with emphasis on diseases involving immune activity. When possible also slight information on the family is registered. Both at the time of admittance and after recovery clinical laboratory tests on somatic status are registered. In addition the level of different cytokines is measured. The psychiatric state and precise diagnoses are registered during the stay. The data will be analysed to uncover connections between psychiatric stress in general as well as specific psychiatric diagnoses and activity in the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the adult acute psychiatric ward of a certain geographical area during the study period

Exclusion Criteria:

* Patients that do not agree to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults aged 18 years and above. Amitted to psychiatric acute ward of St Olavs Hospital, Trondheim, Norway.
Sampling Method: Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
cytokines | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Solveig K Reitan, MD, PhD, Study Chair — St Olavs Hospital/NTNU
Locations (1):
- St Olavs Hospital, Department of Psychiatry, Østmarka Hospital, Trondheim, Middle Norway, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saether SG, Schou M, Stoecker W, Teegen B, Borowski K, Vaaler A, Kondziella D, Reitan SK. Onconeural Antibodies in Acute Psychiatric Inpatient Care. J Neuropsychiatry Clin Neurosci. 2017 Winter;29(1):74-76. doi: 10.1176/appi.neuropsych.16050110. Epub 2016 Aug 31. PMID 27578448
- [Result] Schou M, Saether SG, Borowski K, Teegen B, Kondziella D, Stoecker W, Vaaler A, Reitan SK. Prevalence of serum anti-neuronal autoantibodies in patients admitted to acute psychiatric care. Psychol Med. 2016 Dec;46(16):3303-3313. doi: 10.1017/S0033291716002038. Epub 2016 Sep 9. PMID 27609625
- [Derived] Sakai Y, Iversen V, Reitan SK. FT4 and TSH, relation to diagnoses in an unselected psychiatric acute-ward population, and change during acute psychiatric admission. BMC Psychiatry. 2018 Jul 28;18(1):244. doi: 10.1186/s12888-018-1819-3. PMID 30055589